CLINICAL TRIAL: NCT01335503
Title: Effect of AN-PEP Enzyme on Gastrointestinal Breakdown of Gluten
Brief Title: Effect of AN-PEP Enzyme on Gluten Digestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Food Specialties (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-PEP-02
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Gluten Digestion
Keywords: gluten

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AN-PEP with low caloric meal (Active Comparator)
  Interventions: Dietary Supplement: AN-PEP
- AN-PEP with high caloric meal (Active Comparator)
  Interventions: Dietary Supplement: AN-PEP
- Placebo with low caloric meal (Placebo Comparator)
  Interventions: Dietary Supplement: AN-PEP
- Placebo with high caloric meal (Placebo Comparator)
  Interventions: Dietary Supplement: AN-PEP

INTERVENTIONS:
Dietary Supplement: AN-PEP — Endoprotease enzyme (AN-PEP)
  Other Names: Aspergillus Niger Prolyl EndoProtease enzyme (AN-PEP)

SUMMARY:
The aim is to demonstrate how fast and to what extent AN-PEP can degrade gluten in vivo in the stomach and how much gluten enters the small intestine. A second question is whether the caloric density of a meal can influence the efficacy of AN-PEP breakdown.

DETAILED DESCRIPTION:
In this trial, the effect of AN-PEP enzyme on gastrointestinal breakdown of gluten will be investigated in healthy subjects. In addition, it will be assessed if meal calories can affect the efficacy of AN-PEP. Subjects receive intragastrically, either AN-PEP or placebo, with either a high or a low caloric meal in a double-blind, randomized, placebo-controlled, cross-over fashion. Gastrointestinal fluid will be sampled to measure breakdown of gluten.

ELIGIBILITY:
Inclusion Criteria:

* Male/female
* Age ≥ 18 years but < 45 years
* Hormonal contraceptive treatment
* Subject has read and understood the information provided on the study and given written informed consent

Exclusion Criteria:

* Any medical condition or laboratory test result that in the opinion of the investigators may interfere with the study and may jeopardise the health status of the participant
* pregnancy or lactation
* women not treated with hormonal contraceptive treatment

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Effect of AN-PEP with a low or high caloric meal on gluten degradation in the duodenum | 0-240 min
  Difference in gluten (volume x concentration) x time between AN-PEP and placebo with a low or high caloric meal in the duodenum

SECONDARY OUTCOMES:
Effect of AN-PEP with a low or high caloric meal on gluten degradation in the stomach | 0-240 min
  Difference in gluten concentration x time between AN-PEP and placebo with a low or high caloric meal in the stomach
Effect of meal caloric density on gastric emptying | 0-240 min
  Difference in gastric half emptying time by 13CO2:12CO2 in breath between the high and low caloric meals
Effect of AN-PEP and meal caloric density on gastric and duodenal pH | 0-240 min
  Change in gastric and duodenal pH over time
Effect of caloric density on AN-PEP-mediated gluten degradation in the duodenum | 0-240 min
  Difference in gluten (concentration) x time between AN-PEP with a high vs low caloric meal in the duodenum
Effect of caloric density on AN-PEP-mediated gluten degradation in the stomach | 0-240 min
  Difference in gluten concentration x time between AN-PEP with a high vs low caloric meal in the stomach

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, Prof Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Bartholome R, Salden B, Vrolijk MF, Troost FJ, Masclee A, Bast A, Haenen GR. Paracetamol as a Post Prandial Marker for Gastric Emptying, A Food-Drug Interaction on Absorption. PLoS One. 2015 Sep 9;10(9):e0136618. doi: 10.1371/journal.pone.0136618. eCollection 2015. PMID 26352940
- [Derived] Salden BN, Monserrat V, Troost FJ, Bruins MJ, Edens L, Bartholome R, Haenen GR, Winkens B, Koning F, Masclee AA. Randomised clinical study: Aspergillus niger-derived enzyme digests gluten in the stomach of healthy volunteers. Aliment Pharmacol Ther. 2015 Aug;42(3):273-85. doi: 10.1111/apt.13266. Epub 2015 Jun 4. PMID 26040627